CLINICAL TRIAL: NCT06926504
Title: TeamBirth - an Intervention to Improve Patient Safety and Person-centered Care During Childbirth
Brief Title: TeamBirth-SWE - a Care Process to Improve Safe and Person-centered Intrapartum Care
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University Hospital (Other); Region Skane (Other); Region Halland (Other); Region Jämtland Härjedalen (Other); Ariadne Labs (Other); Värmland County Council, Sweden (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Malin Edqvist, Registered Nurse Midwife, Associate professor, Karolinska Institutet
Other Study IDs: 2023-03517-01; 2024-02476 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2025-03-26; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Person Centered Care; Patient Safety; Patient Satisfaction
Keywords: person-centered care; intrapartum patient safety
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: The care process S-TeamBirth — The intervention consists of the entire care team conducting huddles together with the birthing woman and her partner to plan the care, using the S-TeamBirth whiteboard to communicate and visualize decisions
Behavioral: S-TeamBirth — Involving the entire care team including the woman and her partner in planning the care using team huddles and the S-TeamBirth whiteboard

SUMMARY:
The primary objective of this project is to enhance understanding of intrapartum patient safety and person-centered care through the evaluation of an intervention designed to improve team communication and patient involvement during childbirth, thereby positively impacting maternal and infant health.

Despite various efforts to improve safety in intrapartum care, women and their infants are still harmed. Most adverse events within intrapartum care stem from communication and teamwork failures. Despite national and international recommendations, few interventions target patient safety by incorporating person-centered care.

This project will investigate the effectiveness and implementation of the TeamBirth care process developed by Ariadne Labs Boston, U.S. to improve communication and teamwork among caregivers and women during childbirth. The Swedish version of this care process (TeamBirth-SWE) was adapted, tested, and piloted at Karolinska University Hospital during 2021.

Hypothesis: We hypothesize that the TeamBirth-SWE intervention will have a positive impact on interprofessional teamwork, communication, information sharing, patient involvement, and shared decision-making during labor and birth. These improvements are expected to result in improved maternal and infant outcomes, process measures i.e., patient safety climate, interprofessional collaboration, and improved patient reported measures such as patient involvement, shared-decision-making, and satisfaction with care.

DETAILED DESCRIPTION:
The primary objective of this project is to enhance understanding of intrapartum patient safety and person-centered care through the evaluation of an intervention designed to improve team communication and patient involvement during childbirth, thereby positively impacting maternal and infant health.

Even though childbirth generally is generally considered safe for women in high income countries, the time of birth is critical to the survival of women and their babies, as the risk of morbidity and mortality increases considerably if complications arise. Adverse events reported within maternity care varies from 4-12%, with as much as 57-74% of the incidents being deemed as preventable. According to the Swedish Health and Social Care Inspectorate (IVO), obstetrics and gynecology are one of the areas within somatic specialist care that receive the highest number of complaints. The repercussions of an adverse event or a near miss can have a major impact on both mother and infant, Consequences for women include post-traumatic stress syndrome, secondary fear of birth, and a prolonged interval to a subsequent pregnancy. For infants born with severe asphyxia, the consequences may be lifelong and the societal burden is significant.

Evaluations of teamwork programs or simulation-based teamwork interventions have demonstrated improved team performance and a reduction in morbidity. However, interventions aimed at improving teamwork within intrapartum care have primarily focused on emergency situations, not considering everyday practices. This oversight is significant as many adverse outcomes in intrapartum care develop gradually over time, providing several opportunities for the team to act. Interventions that include person-centered care, facilitate communication and support decision-making processes among interprofessional teams in their daily work have the potential to contribute to enhanced care and outcomes.

The TeamBirth care process was developed by Ariadne Labs, a joint center for health systems innovation at the Harvard T.H Chan School of Public Health (U.S), to improve communication and teamwork between care givers and women to address harmful variation in the quality of intrapartum care. TeamBirth is composed of brief team meetings "huddles" between care givers, women, and their partners, navigated by a shared planning board placed in the birthing room, visible to everyone. The board promotes transparent and reliable communication and includes four areas: (a) the names of the team members, starting with the woman; (b) the woman's preferences; (c) the care plan for the woman, infant, and labor progress; and (d) when the next team huddle is anticipated. TeamBirth has been evaluated for its feasibility and acceptability in the U.S.(25) Given that the intervention has solely been assessed for experiences and implementation, and exclusively within the U.S. context, further research on its effectiveness and whether it functions in other settings is required. We have adapted and tested TeamBirth in the Swedish context in a pilot study conducted at two labor wards in Stockholm during 2022-2023, and the insights have been utilized in the design of the proposed project.

The project addresses the overall aim and the specific research questions in 3 Work Packages (WP):

WP1. Effectiveness of the intervention on patient safety and person-centered care: Does thr TeamBirth-SWE lead to safer care, i.e., improved maternal and infant outcomes during labor, birth and the immediate postnatal period? Will the intervention be more beneficial for women with lower socio-economic status (SES), co-morbidities and high-risk pregnancies?

WP2. Patient reported experiences: Does TeamBirth-SWE improve person-centered care during childbirth? Does it contribute to individualized care, informed choices, shared decision-making, and perceived support from staff?

WP3. Process measures - Patient safety climate and interprofessional collaboration: Does TeamBirth-SWE lead to increased patient safety climate and interprofessional collaboration?

Effectiveness of TeamBirth in reducing adverse maternal and infant outcomes will be evaluated using an interrupted time series design (ITS). The ITS design is particularly suitable for interventions at a population level and over a clearly defined time period, also taking baseline and follow-up trends into account.

WP1. Patient safety outcomes and person-centered care Design, methods: ITS design with segmented regression analysis to study trends in the monthly rates of patient safety outcomes. Data from 2020-2028 will be used; two years before and after implementation at each participating site.

Setting: All labor wards participating in the project Variables/measurements: Patient safety is often measured by composite variables.(30) We decided to choose a primary outcome that reflects the intention of Swedish maternity care: a healthy mother, infant, and a positive experience. In this project we assume that patient involvement and shared decision-making which are cornerstones of person-centered care, contribute to a positive experience. Therefore, two primary outcomes were chosen.

Data sources: Register data from the Swedish Pregnancy Register and the National Swedish Pregnancy Survey 8 weeks after birth (NPS-8). The Swedish Pregnancy Register is a nationwide high-quality register collecting comprehensive data on pregnancy, labor and birth, including maternal health, prenatal care, obstetric interventions, and perinatal outcomes. The Register covers 99% of all births in Sweden and the majority of the variables are retrieved via automatic transfer from the medical record, updated every 24 hours. The NPS-8 is distributed to all pregnant women in gestational week 25, eight weeks and one year after birth. It is available in Swedish, English, Arabic, Farsi, Finnish, French, Spanish, and Somali.

Exposure: The TeamBirth intervention

Primary outcome:

1. Maternal and infant: The composite variable "Birth without major interventions and complications" which, will be used as primary outcome provided from the Swedish Pregnancy Register. It includes the following variables: no operative birth, no postpartum hemorrhage (bleeding>1000 ml), no severe perineal trauma (grade III-IV tears) and a 5-minute Apgar score ≥7.
2. Maternal: NPQ-8 question: "Were you involved in planning and decision-making during birth as much as you wanted to?" (Likert type, scale 1-5)

Secondary outcomes:

1. Maternal: cesarean section, instrumental birth, postpartum hemorrhage (bleeding >1000ml), severe perineal trauma (grade III-IV tears), 8 additional questions reflecting person-centered care from NPQ-8.
2. Infant: 5-minute Apgar score of ≤7, and pH umbilical arterial <7.05.
3. Nine additional questions reflecting person-centered care from the NPS-8.

Covariates: The patient mix before and after the intervention is assumed to be the same. This assumption will be investigated using descriptive time series analysis of potential risk factors for the outcomes, such as the proportion of first-time mothers, smokers, and pre-pregnancy BMI. Furthermore, since the intervention can be started at different times throughout the year, we will adjust for calendar month of birth. High workload, shortage of staff, major organizational changes, or other interventions targeting patient safety are hypothesized to be potential confounders. To account for high-workload, we will use the number of births per 24 hours. Another possible confounder is major long-term disturbances in the work situation, which will be addressed in sensitivity analyses, where a priori defined time periods of follow-up will be excluded, i.e., based on known periods of organizational turbulence, shortage of midwives, or other major changes.

Power calculation: In 2020, approximately 80% of the births at the study sites were without major interventions or complications, with 51% of women being completely satisfied with their participation in decision-making. Based on observed standard deviations from 2020, we estimate this study has 80% power (at 5% significance with a 2-sided test) to detect a 1.3 percent point increase in the proportion of births without major adverse events and a 2.5% percent point increase in the proportion of women completely satisfied with their participation during labor and birth. The latter outcome is measured on a Likert scale, and an analysis of ordinal data is expected to further increase statistical power. Since the intervention is complex, our hypothesis is a successive improvement of 1.5 percentage points each year for "births without major interventions and complications", and by 5 percentage points per year for the variable "satisfied with participation in decision-making".

Analysis: The proportion of women with the defined outcomes, per calendar month and study site, will be analyzed using multiple regression, weighted proportionally to the number of pregnancies per month. The basic model will include study site, calendar month, and a time variable divided into pre-intervention, 0-6 months, and 7-18 months after implementation. If trends in outcomes before the intervention are observed, analyses based on change of trends before and after intervention will also be performed. As the effect of the intervention may vary by population characteristics, we will perform stratified analyses based on parity, onset of labor, and study site.

WP2. Patient reported experience measures Design, methods: A web-based survey, including background questions, validated scales and study specific items, will be sent to women one month after birth. The survey will be available in Swedish and English.

Inclusion criteria: All women >15 years of age with spontaneous onset of labor or induction of labor after gw 22+0, and who are proficient in Swedish or English.

Exclusion criteria: Planned caesarean section, intrauterine fetal demise. Instruments: Validated scales will be used; Mothers Autonomy in Decision-making (MADM), Mothers on Respect Index (MOR), Mistreatment Index (MIST) and Childbirth Experience Questionnaire 2.0 (CEQ2) and Support and Control in Birth Scale (SCIB). Women will be asked about their experience of S-TeamBirth during their labor and birth.

Exposure: Women experiencing high use of TeamBirth-SWE (>5 huddles). Outcome: Primary outcome: Women's experiences of autonomy and shared decision-making (MADM). Secondary outcomes: Mothers on Respect Index (MOR), the Mistreatment Index (MIST), the Childbirth Experience questionnaire (CEQ2) and the Support and Control in Birth Scale (SCIB).

Exploratory factors: Mode of birth, adverse maternal or neonatal outcomes, fear of birth. Any imbalances between the groups related to background and pregnancy characteristics will be accounted for.

WP3. Patient safety climate and interprofessional collaboration Design, methods: A longitudinal cross-sectional design, using survey data measured at four time points.

Participants: All midwives, physicians and nurse assistants working with intrapartum care at the participating labor wards.

Instruments and measurements: Validated scales will be used; The Hospital Survey on Patent Safety (HSPOS 2.0) to measure patient safety climate and the Assessment of Collaborative Environments (ACE-15) to conceptualize the dimensions of interprofessional teamwork. Timepoints for measurement: One month before the start of the implementation (T0), 6 months (T1), 12 months (T2), and 24 months (T3) after the implementation of S-TeamBirth.

To assess the effect of TeamBirth-SWE on patient safety climate and interprofessional teamwork, data from pre- and post-intervention will be compared. Furthermore, the effect of the intervention will be analyzed over time. Data normality will be tested using the Shapiro-Wilk test, and ANOVA with repeated measures or Friedman's test will be conducted to compare the mean scores (dimensions and total scores) and assess differences between the time points (T0-T3). Posthoc tests will be performed to investigate differences in attitudes between professions. Differences in mean change scores will further be calculated for three samples to assess when (or if) changes in attitudes occur: Sample 1 (T1 compared to T0), Sample 2 (T2 compared to T1), and Sample 3 (T3 compared to T1) using t-tests or Mann-Whitney U-tests. If samples are proven to be dependent, a paired t-test or Wilcoxon signed-rank test will be employed.

ELIGIBILITY:
Inclusion criteria:

* Spontaneous onset of labor
* Induction of labort
* Gestational week >22+0

Exclusion criteria:

* Planned cesarean section
* Intrauterine Fetal Demise
* Gestational week <22+0, .

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consist of all women who fulfill the inclusion criteria at the participating labor wards.
Sampling Method: Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2028-09-05 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth without major interventions or complications | From labor ward admission to discharge home, to 4 hours postpartum.
  The primary outcome is a composite measure including provided by the Swedish Pregnancy register and includes the following variables: no operative birth, no postpartum haemorrhage (>1000 ml), no severe perineal trauma, and a 5-minute Apgar score >=7.
Shared intrapartum decision-making | PREM data collected 8 weeks after birth
  Were you involved in planning and decision-making to your desired extent? Likert type question in the Swedish National Pregnancy Survey

SECONDARY OUTCOMES:
Unplanned cesarean section | At delivery/birth
  Mode of birth; caesarean section
Spontaneous vaginal birth | From labour onset to birth of the baby
  Mode of birth, spontaneous
Instrumental birth | From labour onset to instrumental birth performed
  Mode of birth, vacuum extraction/forceps
Postpartum bleeding | From brith of the baby to 4 hours after birth
  Postpartum bleeding in ml, >500 ml, >1000 ml
Severe perineal trauma | Diagnosed at birth to 24 hours after birth
  Injuries affecting the anal sphincter O70.2, O70.3
Apgar score <7 at 5 minutes | Measured at 5 minutes after birth
  Apgar score less than 7 at 5 minutes after birth
Apgar score <4 at 5 minutes | Measured at 5 minutes after birth
  Apgar score less than 4 at 5 minutes after birth
Umbilical arterial pH | From birth to 20 minutes after birth
  pH measured from the umbilical artery at birth
Adequeate pain relief | PREM data collected 8 weeks after birth
  Did you receive adequate pain relief during childbirth? Likert type question in the Swedish National Pregnancy Survey
Support from staff | PREM data collected 8 weeks after birth
  Did you receive support from the staff during your delivery to the extent you desired? Likert type question in the Swedish National Pregnancy Survey
Midwifery presence during childbirth | PREM data collected 8 weeks after birth
  Was the midwife present in the birthing room to the extent you desired? Likert type question in the Swedish National Pregnancy Survey
Staff collaboration | PREM data collected 8 weeks after birth
  Did the staff collaborate effectively? Likert type question in the Swedish National Pregnancy Survey
Respectful care | PREM data collected 8 weeks after birth
  Were you treated with respect during labour and birth? Likert type question in the Swedish National Pregnancy Survey
Sufficient information | PREM data collected 8 weeks after birth
  Did you receive sufficient information during childbirth? Likert type question in the Swedish National Pregnancy Survey
Safe care | PREM data collected 8 weeks after birth
  Did you feel safe with the care provided during childbirth? Likert type question in the Swedish National Pregnancy Survey
Partner's involvement during childbirth | PREM data collected 8 weeks after birth
  Did the staff involve your partner/relative to the extent you desired? Likert type question in the Swedish National Pregnancy Survey
Women's experience of autonomy in decision-making during childbirth | Questionnaire sent to women 4 weeks after birth
  Mothers Autonomy in Decision-making (MADM) scale. 7 questions, rated on a six point Likert scale from Strongly Disagree to Strongly Agree.
Women's experience of respect during childbirth | Questionnaire sent to women 4 weeks after birth
  Measure of Respect Index (MOR). 14 items, rated on a 6-point Likert scale
Women's overall childbirth experience | Questionnaire sent to women 4 weeks after birth
  Childbirth Experience Questionnaire 2.0 (CEQ2): 22 items rated on a 4-point Likert scale from Totally Disagree to Totally Agree.
Women's experience of mistreatment during childbirth | Questionnaire sent to women 4 weeks after birth
  The Mistreatment Index (MIST). 7 items, yes/no response
Women's experience of support and control during childbirth | Questionnaire sent to women 4 weeks after birth
  SCIB: 33 items rated on a 5-point Likert scale from Agree Completely to Disagree Completely.
Patient safety climate | Longitudinal questionnaire sent to all staff working with intrapartum care at the participating study sites, measured at baseline before study start, 6 months, 12, monts and 24 months after study start
  The Hospital Survey on Patent Safety Culture (HSPOS 2.0) 40 items rated on a 5-point Likert scale from Strongly Disagree to Strongly Agree plus an additional response; Not applicable
Interprofessional teamwork | Longitudinal questionnaire sent to all staff working with intrapartum care at the participating study sites, measured at baseline before study start, 6 months, 12, monts and 24 months after study start
  Interprofessional teamwork will be measured using the Assessment of Colloborative Environments scale (ACE-15)

CONTACTS AND LOCATIONS:
Locations (7):
- Sweden (7):
  - Region Halland, labour ward Halmstad, Halmstad Hospital, Halmstad, Halland County
  - Region Halland, labour ward Varberg County Hospital, Varberg, Halland County
  - Department of Women's Health, Labour ward Östersund County Hospital, Östersund, Region Jämtland Härjedalen
  - Region Skåne, labour wards Lund & Malmö, Lund, Skåne County
  - Department of Women's Health, labour ward Uppsala University Hospital, Uppsala, Uppsala County
  - Department of Women's Health, Labour ward Karlstad County Hospital, Karlstad, Värmland County
  - Department of Women's Health, Labour ward Solna & Huddinge, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
The data might be shared after discussions with researchers who apply to the Swedish Ethical Review Authorities and with data sharing agreements in place.

REFERENCES:
- [Background] Aibar L, Rabanaque MJ, Aibar C, Aranaz JM, Mozas J. Patient safety and adverse events related with obstetric care. Arch Gynecol Obstet. 2015 Apr;291(4):825-30. doi: 10.1007/s00404-014-3474-3. Epub 2014 Sep 23. PMID 25245667
- [Background] Skoogh A, Hall-Lord ML, Baath C, Bojo AS. Adverse events in women giving birth in a labor ward: a retrospective record review study. BMC Health Serv Res. 2021 Oct 14;21(1):1093. doi: 10.1186/s12913-021-07109-5. PMID 34649538
- [Background] Dencker A, Nilsson C, Begley C, Jangsten E, Mollberg M, Patel H, Wigert H, Hessman E, Sjoblom H, Sparud-Lundin C. Causes and outcomes in studies of fear of childbirth: A systematic review. Women Birth. 2019 Apr;32(2):99-111. doi: 10.1016/j.wombi.2018.07.004. Epub 2018 Aug 14. PMID 30115515
- [Background] Hill MG, Reed KL, Brown RN; Newborn Brain Society Guidelines and Publications Committee. Perinatal asphyxia from the obstetric standpoint. Semin Fetal Neonatal Med. 2021 Aug;26(4):101259. doi: 10.1016/j.siny.2021.101259. Epub 2021 Jun 11. PMID 34175240
- [Background] Kurinczuk JJ, White-Koning M, Badawi N. Epidemiology of neonatal encephalopathy and hypoxic-ischaemic encephalopathy. Early Hum Dev. 2010 Jun;86(6):329-38. doi: 10.1016/j.earlhumdev.2010.05.010. Epub 2010 Jun 16. PMID 20554402
- [Background] Wu M, Tang J, Etherington C, Walker M, Boet S. Interventions for improving teamwork in intrapartem care: a systematic review of randomised controlled trials. BMJ Qual Saf. 2020 Jan;29(1):77-85. doi: 10.1136/bmjqs-2019-009689. Epub 2019 Oct 10. PMID 31601734
- [Background] Liberati EG, Tarrant C, Willars J, Draycott T, Winter C, Kuberska K, Paton A, Marjanovic S, Leach B, Lichten C, Hocking L, Ball S, Dixon-Woods M; SCALING Authorship Group. Seven features of safety in maternity units: a framework based on multisite ethnography and stakeholder consultation. BMJ Qual Saf. 2021 Jun;30(6):444-456. doi: 10.1136/bmjqs-2020-010988. Epub 2020 Sep 25. PMID 32978322
- [Background] Aggarwal R, Plough A, Henrich N, Galvin G, Rucker A, Barnes C, Berry W, Golen T, Shah NT. The design of "TeamBirth": A care process to improve communication and teamwork during labor. Birth. 2021 Dec;48(4):534-540. doi: 10.1111/birt.12566. Epub 2021 Jul 9. PMID 34245054
- [Background] Weiseth A, Plough A, Aggarwal R, Galvin G, Rucker A, Henrich N, Miller K, Subramanian L, Hawrusik R, Berry W, Gullo S, Spigel L, Dever K, Loveless D, Graham K, Paek B, Shah NT. Improving communication and teamwork during labor: A feasibility, acceptability, and safety study. Birth. 2022 Dec;49(4):637-647. doi: 10.1111/birt.12630. Epub 2022 Mar 1. PMID 35233810
- [Background] Neergheen VL, Chaer LE, Plough A, Curtis E, Paterson VJ, Short T, Bright A, Lipsitz S, Murphy A, Miller K, Subramanian L, Radichel E, Ervin J, Castleman L, Brown E, Yeboah T, Simas TM, Terk D, Vedam S, Shah N, Weiseth A. Assessing patient autonomy in the context of TeamBirth, a quality improvement intervention to improve shared decision-making during labor and birth. Birth. 2024 Dec;51(4):855-866. doi: 10.1111/birt.12857. Epub 2024 Aug 14. PMID 39140579
- [Background] Bernal JL, Cummins S, Gasparrini A. Interrupted time series regression for the evaluation of public health interventions: a tutorial. Int J Epidemiol. 2017 Feb 1;46(1):348-355. doi: 10.1093/ije/dyw098. PMID 27283160
- [Background] Vedam S, Stoll K, Rubashkin N, Martin K, Miller-Vedam Z, Hayes-Klein H, Jolicoeur G; CCinBC Steering Council. The Mothers on Respect (MOR) index: measuring quality, safety, and human rights in childbirth. SSM Popul Health. 2017 Jan 19;3:201-210. doi: 10.1016/j.ssmph.2017.01.005. eCollection 2017 Dec. PMID 29349217
- [Background] Vedam S, Stoll K, Taiwo TK, Rubashkin N, Cheyney M, Strauss N, McLemore M, Cadena M, Nethery E, Rushton E, Schummers L, Declercq E; GVtM-US Steering Council. The Giving Voice to Mothers study: inequity and mistreatment during pregnancy and childbirth in the United States. Reprod Health. 2019 Jun 11;16(1):77. doi: 10.1186/s12978-019-0729-2. PMID 31182118
- [Background] Walker KF, Dencker A, Thornton JG. Childbirth experience questionnaire 2: Validating its use in the United Kingdom. Eur J Obstet Gynecol Reprod Biol X. 2019 Oct 3;5:100097. doi: 10.1016/j.eurox.2019.100097. eCollection 2020 Jan. PMID 32021972
- [Background] Waterson P, Carman EM, Manser T, Hammer A. Hospital Survey on Patient Safety Culture (HSPSC): a systematic review of the psychometric properties of 62 international studies. BMJ Open. 2019 Sep 4;9(9):e026896. doi: 10.1136/bmjopen-2018-026896. PMID 31488465
- [Background] Tilden VP, Eckstrom E, Dieckmann NF. Development of the assessment for collaborative environments (ACE-15): A tool to measure perceptions of interprofessional "teamness". J Interprof Care. 2016 May;30(3):288-94. doi: 10.3109/13561820.2015.1137891. Epub 2016 Mar 30. PMID 27029641
- [Background] Ford E, Ayers S, Wright DB. Measurement of maternal perceptions of support and control in birth (SCIB). J Womens Health (Larchmt). 2009 Feb;18(2):245-52. doi: 10.1089/jwh.2008.0882. PMID 19183096